CLINICAL TRIAL: NCT04889170
Title: Prevalence of Subclinical and Clinical Dysphagia in Parkinson's Disease and Evaluation of the NRZ Dysphagia Pathway
Brief Title: Prevalence of Subclinical and Clinical Dysphagia in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Neurological Rehabilitation Hospital Rosenhügel (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Other Study IDs: NRZ_EK-20-135-0820
Record Dates: First submitted 2021-04-26; First posted 2021-05-17 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease; Dysphagia
Keywords: FEES
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biofeedback therapy + Voice training: The intervention has two parts. One part of the intervention is the biofeedback therapy. The biofeedback therapy means that the patient and a speech and language therapist watch the video of the FEES together and discuss the findings. The other part of the intervention is a voice training. The frequency of therapy is minimum 3 times a week, the duration of one therapy is minimum 25 minutes.
  Interventions: Other: Intervention
- Biofeedback therapy + Swallow training: The intervention has two parts. One part of the intervention is the biofeedback therapy. The biofeedback therapy means that the patient and a speech and language therapist watch the video of the FEES together and discuss the findings. The other part of the intervention is a swallow training. The frequency of therapy is minimum 3 times a week, the duration of one therapy is minimum 25 minutes.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Intervention: After recording the patient characteristics and the baseline dysphagia characteristics, the intervention begins. The intervention lasts 3 weeks, by extended stay it lasts 5 or 7 weeks.
  The intervention has two parts. One part of the intervention is the biofeedback therapy. The biofeedback therapy means that the patient and an SLT watch the video of the FEES together and discuss the findings. The other part of the intervention is a swallow training or a voice training. The frequency of therapy is minimum 3 times a week, the duration of one therapy is minimum 25 minutes.
  Allocation to the Groups will be done by a randomization software

SUMMARY:
Background:

In idiopathic Parkinson's disease, 50% of patients develop in the course of the disease a dysphagia and aspiration pneumonia is the leading cause of death in all parkinsonian syndromes . Dysphagia can negatively impact on the course of Parkinson's disease due to complications such as aspiration pneumonia, malnutrition, inadequate drug action, it causes a deterioration in quality of life and leads to an increase in health care costs of more than 10% Therefore, it is very important to detect subclinical dysphagia in time in Parkinson's disease and to initiate a targeted swallowing therapy. In the Neurological Rehabilitation Center Rosenhügel, patients with Parkinson's disease participate in the Parkinson rehabilitation pathway during their rehabilitation program. A part of the Parkinson rehabilitation pathway is the dysphagia pathway. It includes a clinical swallowing examination, an instrumental assessment of swallowing, performed by a fiberoptic endoscopic evaluation of swallowing (FEES) and a dysphagia training. Because of the serious clinical consequences of dysphagia, the investigators decided to further evaluate the prevalence of subclinical and clinical dysphagia in Parkinson's disease and to assess the efficacy of the NRZ dysphagia pathway. Our goal is to detect and classify all Parkinson's disease patients with dysphagia and to prevent the complications of dysphagia by an early therapeutic intervention.

Objectives Primary objective: Evaluation of prevalence of dysphagia in Parkinson's disease Secondary objective: Evaluation of the impact of the NRZ dysphagia pathway on the severity of dysphagia through vocal training or dysphagia training Methods A prospective cohort study will be conducted for 24 months. All patients with the diagnosis of a Parkinson's disease, who are treated as inpatients in the Neurological Rehabilitation Center Rosenhügel from 5/2020 till 5/2022 and have signed an informed consent form will be enrolled in the study. The patients will be examined for dysphagia by a clinical swallowing examination, by a FEES and by measuring the swallowing related quality of life before and after dysphagia training.

Intervention A dysphagia training, which consists of a biofeedback therapy and a swallow training or a voice training. The intervention lasts 3 weeks, by extended stay it lasts 5 or 7 weeks.

DETAILED DESCRIPTION:
Background:

In idiopathic Parkinson's disease, 50% of patients develop in the course of the disease a dysphagia and aspiration pneumonia is the leading cause of death in all parkinsonian syndromes. Dysphagia in idiopathic Parkinson's disease is subjectively perceived and communicated only in the late stages. Dysphagia can negatively impact on the course of Parkinson's disease due to complications such as aspiration pneumonia, malnutrition, inadequate drug action, it causes a deterioration in quality of life and leads to an increase in health care costs of more than 10% . Therefore, it is very important to detect subclinical dysphagia in time in Parkinson's disease and to initiate a targeted swallowing therapy. Simple screening methods are insufficient for the diagnosis of subclinical swallowing disorders. In the Neurological Rehabilitation Center Rosenhügel, patients with Parkinson's disease participate in the Parkinson rehabilitation pathway during their rehabilitation program. A part of the Parkinson rehabilitation pathway is the dysphagia pathway. It includes a clinical swallowing examination, an instrumental assessment of swallowing, performed by a fiberoptic endoscopic evaluation of swallowing (FEES) and a dysphagia training. Because of the serious clinical consequences of dysphagia, the investigators decided to further evaluate the prevalence of subclinical and clinical dysphagia in Parkinson's disease and to assess the efficacy of the NRZ dysphagia pathway. Our goal is to detect and classify all Parkinson's disease patients with dysphagia and to prevent the complications of dysphagia by an early therapeutic intervention.

Objectives Primary objective: Evaluation of prevalence of dysphagia in Parkinson's disease Secondary objective: Evaluation of the impact of the NRZ dysphagia pathway on the severity of dysphagia through vocal training or dysphagia training Methods A prospective cohort study will be conducted for 24 months. All patients with the diagnosis of a Parkinson's disease, who are treated as inpatients in the Neurological Rehabilitation Center Rosenhügel from 5/2020 till 5/2022 and have signed an informed consent form will be enrolled in the study. The patients will be examined for dysphagia by a clinical swallowing examination, by a FEES and by measuring the swallowing related quality of life before and after dysphagia training.

Intervention A dysphagia training, which consists of a biofeedback therapy and a swallow training or a voice training. The intervention lasts 3 weeks, by extended stay it lasts 5 or 7 weeks.

Results The primary endpoint is the prevalence of clinical and subclinical dysphagia in patients with Parkinsons'disease. Secondary endpoints are the change in the food texture modification categorie as well as the changes in the liquid texture modification categorie, in the Rosenbek Penetration-Aspiration Scale, in the drooling scale an in the swallowing-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a Parkinson's disease
* Inpatient in the Neurological Rehabilitation Center Rosenhügel from 12/2020 till 12/2022
* Informed consent form signed

Exclusion Criteria:

* General contraindications of fiberoptic endoscopic evaluation of swallowing.
* Not feasible fiberoptic endoscopic evaluation of swallowing due to anatomical changes.
* Not feasible fiberoptic endoscopic evaluation of swallowing due to hypersensitivity .
* Not feasible fiberoptic endoscopic evaluation of swallowing due to incompliance.
* Pregnancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of a Parkinson's disease, who are treated as inpatient in the Neurological Rehabilitation Center Rosenhügel from 12/2020 till 12/2022 and have signed an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of dysphagia | 24 Months
  Primary objectives (Hypothesis): Evaluation of prevalence of dysphagia in Parkinson's disease. We assume that 30 percent of the patients will have a clinical dysphagia and 70 percent will have no clinical dysphagia.

SECONDARY OUTCOMES:
Evaluation of the impact of the NRZ dysphagia pathway on the severity of dysphagia as measured by the Rosenbek Penetration-Aspiration Scale | 24 Months
  Description oft he Rosenbek Penetration Aspiration Scale The Rosenbek Penetration Aspiration Scale is an eight point scale, which ranks the two cardinal dysphagia symptoms, penetration and aspiration. The values 2-5 correspond to a penetration and 6-8 to an aspiration. Minimum value: 1 point, maximum value: 8 points; higher scores mean a worse outcome.
Evaluation of the impact of the NRZ dysphagia pathway on the severity of dysphagia as measured by the food texture modification categorie | 24 Months
  There are 7 categories for food texture modification:
  Category 1: normal diet (Score: 1 Point) Category 2: Individual phase diet (Score: 2 Points) Category 3: Phase 4 (semi-soft and solid food that can be easily chewed) (Score: 3 Points) Category 4: Phase 3 (softly cooked, easy to mash with the tongue on the palate) (Score: 4 Points) Category 5: Phase 2 (soups/sauces/dessert/breakfast mushy/homogeneous) (Score: 5 Points) Category 6: Phase 1 (all foods mushy/homogenous) (Score: 6 Points) Category 7: Phase 0 (no oral food intake possible) (Score: 7 Points) Minimum value: 1 point, maximum value: 7 points; higher scores mean a worse outcome.
Evaluation of the impact of the NRZ dysphagia pathway on the severity of dysphagia as measured by the liquid texture modification categorie | 24 Months
  There are 8 categories for liquid texture modification:
  Category 1: Nonthickened liquid (Score: 1 Point) Category 2: 0.5 MB/200ml thickened liquid (Score: 2 Points) Category 3: 1 MB/200ml thickened liquid (Score: 3 Points) Category 4: 1.5 MB/200ml thickened liquid (Score: 4 Points) Category 5: 2 MB/200ml thickened liquid (Score: 5 Points) Category 6: 2,5 MB/200ml thickened liquid (Score: 6 Points) Category 7: 3 MB/200ml thickened liquid (Score: 7 Points) Category 8: no oral fluid intake possible (Score: 8 Points) Minimum value: 1 point, maximum value: 8 points; higher scores mean a worse outcome.
Evaluation of the impact of the NRZ dysphagia pathway on the severity of dysphagia as measured by the Drooling Severity and Frequency Scale | 24 Months
  Description of the Drooling Severity and Frequency Scale Frequency and spatial extent are recorded. The two individual values together give a total value between 2 (never) and 9. Minimum value: 2 points, maximum value: 9 points; higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurological Rehabilitation Center Rosenhügel, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No